CLINICAL TRIAL: NCT03385954
Title: Effectiveness of a Distance Eduaction Course for Prevention in RSI/WRMD on Life Quality of a Nursing Group
Brief Title: Effectiveness of a Distance Eduaction Course for Prevention in RSI/WRMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160415
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-10

CONDITIONS: Work-related Injury
Keywords: nursing; distance; education; RSI/WRMD
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): distance education curse with 8 hours to be accomplished in 2 weeks,
  Interventions: Other: Intervention
- Control (Experimental): Wiil receive a lecture of 30 minutes
  Interventions: Other: Control

INTERVENTIONS:
Other: Intervention — The distance eduacation group course has a workload of 8 hours and will be developed over 2 weeks. It is suggested that students have a minimum of 1 hour of study per day. The course will consist of work tips, clarifications and procedures for the prevention of RIS/WRMD physical training tips to improve cardiovascular condition and, of strength and flexibility, available literature and theoretical evidence that should be answered through the knowledge acquired in the EAD course of prevention of LERDORT from the HCPA's Physiatrics and Rehabilitation Service. This Course will be available through moodle.
  Arms: Intervention
Other: Control — will receive a lecture of 30 minutes.
  Arms: Control

SUMMARY:
Repetitive Strain Injuries (RSI) or Work-Related Ostomuscular Disorders (WRMD) are musculoskeletal disorders. Nursing is one of the categories of workers most affected, due to the inherent functions they perform in their daily activities. The objective of this study is to evaluate the effects of a distance education program of prevention in RIS/WRMD on the quality of life of a nursing group.

DETAILED DESCRIPTION:
Repetitive Strain Injury (RSI) or Work-Related Musculoskeletaldisorders (WRMD) are the names given to skeletal muscle disorders that mainly affect the upper limbs, the scapular region and the neck. One of the most affected categories is nursing workers who present health problems inherent to the function they perform in their daily activities. Due to this peculiarity, several studies are focused on the occupational risks of nursing workers in the hospital environment. However, It was not found in the literature studies that suggests strategies to prevent and improve the worker's quality of life. Distance education comes as a differential. It has power in interactive media and collaborative learning beyond self-learning and mass media. This research project proposes to carry out a randomized clinical trial where the intervention group will receive a Prevention Course in RSI/WRMD in the distance education modality and the control group will receive Educational Lectures on Prevention in RSI /WRMD, both groups will be composed by a nursing team from the Clinical Hospital of Porto Alegre.

ELIGIBILITY:
Inclusion Criteria:

* Nurse staff from HCPA
* Male and Female
* Individuals that agree to participate of the distance eduacational course
* Individuals that agree to participate in the research by signing the Term of Free and Clarified Consent

Exclusion Criteria:

* Individuals that do not complete the course
* Individuals that do not agree to participate in the research by signing the Term of Free and Clarified Consent
* Individuals with chronic musculoskeletal injury diagnosed.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-03-30 (Estimated); Study Completion 2019-03-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 48 months
  Verified by instrument SF36 - With 36 items that measure eight domains (variables): functional capacity, physical aspects, pain, general health, vitality, social aspects, emotional aspects and mental health. The highest score for each SF-36 domain is 100 and the lowest score is 0.

CONTACTS AND LOCATIONS:
Overall Officials: Antônio C dos Santos, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Pôrto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Corlett EN, Bishop RP. A technique for assessing postural discomfort. Ergonomics. 1976 Mar;19(2):175-82. doi: 10.1080/00140137608931530. No abstract available. PMID 1278144
- [Background] Lincoln AE, Feuerstein M, Shaw WS, Miller VI. Impact of case manager training on worksite accommodations in workers' compensation claimants with upper extremity disorders. J Occup Environ Med. 2002 Mar;44(3):237-45. doi: 10.1097/00043764-200203000-00011. PMID 11911025